CLINICAL TRIAL: NCT04084262
Title: Correction of Multi-Plane Hallux Valgus Deformity Using the Phantom® Intramedullary Nail
Brief Title: Multi-Plane Hallux Valgus Correction With the Phantom® Nail
Status: Completed | Type: Observational
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P30-SP-0002
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Arthrodesis; Bunion; Hallux Valgus
Keywords: bunion; supinating reduction; multi-plane; lapidus; arthrodesis; intramedullary nail; hallux valgus
MeSH Terms: conditions — Ankylosis; Bunion; Hallux Valgus | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Study Participants: Phantom® Intramedullary Nail combined with a supinating reduction technique
  Interventions: Device: Intramedullary Nail

INTERVENTIONS:
Device: Intramedullary Nail — Subjects undergo a Lapidus Arthrodesis procedure combined with a supinating reduction technique to create a multi-plane correction of hallux valgus
  Other Names: Phantom® Intramedullary Nail

SUMMARY:
The goal of this research study is to determine the change in frontal plane rotation of the 1st metatarsal from pre to post arthrodesis of the 1st TMT joint with the Phantom® Intramedullary Nail combined with a supinating reduction technique.

The study hypothesis is that multi-planar correction can be achieved with the Phantom® Intramedullary Nail.

DETAILED DESCRIPTION:
Each subject will undergo a Lapidus Arthrodesis combined with a supinating reduction technique.

The subjects will undergo 3 weight-bearing CBCT scans of their foot and ankle, one pre-arthrodesis, one two weeks post-arthrodesis, and one 12 weeks post-arthrodesis. These scans will be used to determine change in frontal plane rotation of the 1st metatarsal from pre to post arthrodesis of the 1st TMT joint, change in angular/positional alignment of the 1st TMT joint using various measurements (1-2 IMA, Meary's Angle, HVA, MAA, Sesamoid Position, and Sesamoid Frontal Plane Rotation), maintenance of correction of the 1st TMT joint, and union status.

The subjects will also complete three surveys, the Pain and Satisfaction Survey, the AOFAS Hallux MTP-IP Scale, and the FAOS Foot and Ankle Survey, at the Pre-Operative Visit, 2 Week Visit (post-op), 6 Week Visit (post-op), and 12 Week Visit (post-op). Furthermore, the subjects will be asked about their willingness to undergo the procedure again at the 12 Week Visit (post-op). All of these scores will be considered in the secondary objectives.

Aside from the study activities listed above, all procedures, visits, and instructions for the subject are to follow the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age at the time of screening.
* The subject has been diagnosed with hallux valgus.
* The subject has pain associated with hallux valgus.
* The subject agrees to comply with the requirements of the study and complete the study measures.
* The subject is willing and able to provide written informed consent.
* The subject plans to undergo a Lapidus Arthrodesis procedure with a 3-Hole Phantom® Intramedullary Nail.

Exclusion Criteria:

* The subject is pregnant.
* The subject has had previous surgery for hallux valgus on operative side.
* The subject will require a structural graft in the 1st TMT joint.
* The unshod foot in question is greater than 28 cm in length.
* The subject is not expected to complete the study according to the investigation plan.
* The subject has been deemed physiologically or psychologically inadequate by the enrolling physician.
* The subject is a prisoner, unable to understand what participation in the study entails, mentally incompetent, a known abuser of alcohol and/or drugs, or anticipated to be non-compliant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults age 18 and older with a hallux valgus deformity. The most common age demographic to have surgery for hallux valgus correction is age 50-59. Additionally, the prevalence of hallux valgus in females is greater than males, so a higher percentage of female subjects seeking treatment is likely to be expected.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Frontal Plane Rotation | 12 weeks
  Determine the change in frontal plane rotation of the 1st metatarsal from pre to post arthrodesis of the 1st tarsometatarsal joint with the Phantom® Intramedullary Nail combined with a supinating reduction technique.

SECONDARY OUTCOMES:
1-2 Inter Metatarsal Angle | Pre-op, 2 weeks, 12 weeks
  Change in 1-2 Inter Metatarsal Angle before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Meary's Angle | Pre-op, 2 weeks, 12 weeks
  Change in Meary's Angle before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Hallux Valgus Angle | Pre-op, 2 weeks, 12 weeks
  Change in Hallux Valgus Angle before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Metatarsus Adductus Angle | Pre-op, 2 weeks, 12 weeks
  Change in Metatarsus Adductus Angle before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Sesamoid Position | Pre-op, 2 weeks, 12 weeks
  Change in sesamoid position before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Sesamoid Frontal Plane Rotation | Pre-op, 2 weeks, 12 weeks
  Change in sesamoid frontal plane rotation before and after arthrodesis of the 1st tarsometatarsal joint using weightbearing CBCT imaging
Maintenance of Correction | Pre-op, 2 weeks, 12 weeks
  Maintenance of lapidus arthrodesis correction via CBCT analysis
Union Status | 12 weeks
  Union/delayed union status at 12 Week Visit
Clinical Complications | Pre-Op, 2 weeks, 6 weeks,12 weeks
  Any lapidus arthrodesis related clinical complications
Patient Current Level of Pain at Surgical Site | Pre-Op, 2 weeks, 6 weeks, 12 weeks
  Visual Analog Scale (VAS). Line from 0 (no pain) to 10 (worst pain). Patient reported.
AOFAS | Pre-Op, 2 weeks, 6 weeks, 12 weeks
  Change in AOFAS Hallux Metatarsophalangeal-Interphalangeal Scale scores
  AOFAS Hallux Metatarsophalangeal-Interphalangeal Scale foot clinical score. Pain: 0-40 points Function: 0-45 points Alignment: 0-15 points Total Score (sum): 0-100 points (higher score indicates better outcomes)
FAOS | Pre-Op, 2 weeks, 6 weeks, 12 weeks
  Change in FAOS Foot and Ankle Survey scores
  Standardized answer options are given (% Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
  Subscales:
  Pain Other Symptoms Functions in Daily Living (ADL) Function in sport and recreation Foot and ankle-related Quality of Life (QoL)
Patient Satisfaction with Procedure | Pre-Op, 2 weeks, 6 weeks, 12 weeks
  Patient reported satisfaction by check boxes (Likert Scale) from Pain and Satisfaction Survey
Willingness to Undergo Procedure Again | 12 weeks
  Willingness to undergo procedure again (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Brinker, DPM, Study Director — Director of Clinical Research
Locations (1):
- Orthopedic Center of Palm Beach County, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No